CLINICAL TRIAL: NCT04023799
Title: Dual Purpose Prevention (DPP) Product Preferences Among Couples
Brief Title: Couple User Preferences in Dual Purpose Prevention Products
Acronym: CUPID
Status: Completed | Type: Observational
Sponsor: Microbicide Trials Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: MTN-045; UM1AI068633 (NIH); UM1AI068615 (NIH); UM1AI106707 (NIH); 38598 (Other: DAIDS)
Record Dates: First submitted 2019-03-14; First posted 2019-07-18 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: HIV Prevention; Contraception Behavior
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
MTN-045 is a cross-sectional study that will utilize questionnaires, including Discrete-Choice Experiments (DCE) and joint decision tasks, to assess couples' preferences related to dual purpose prevention (DPP) products that could be used to prevent unintended pregnancies and HIV infection. Post-survey explanatory in-depth interviews (IDIs) will be conducted with a subset of participants to explore DPP product-related decisions..

DETAILED DESCRIPTION:
MTN-045 is a cross-sectional study that will utilize questionnaires, including DCEs and joint decision tasks, and IDIs to assess heterosexual couples' preferences related to DPP products that could be used to prevent unintended pregnancies and HIV infection. One main goal of the study is to determine heterosexual couples' preferences for a DPP product to inform product delivery and future product design to maximize uptake and willingness to use among sub-Saharan African heterosexual couples. Another main goal of the study is to assess the level of influence of the male partner on a woman's preferences for a DPP product and on her decision-making process regarding product preferences and use.

The MTN-045 study population will consist of approximately 400 heterosexual sub-Saharan African couples of reproductive age who have been in a relationship for ≥ 3 months and are interested in contraception and/or HIV prevention. Women who are currently using contraceptives as well as those not using contraceptives will be eligible. Couples who are living together as well as those not living together will be eligible. All participants will complete survey questionnaires, first separately from their partner, then followed by a joint couples' decision task. Up to 80 participants, i.e., one or both partners from a subset of up to 40 couples, will be selected to complete an IDI.

ELIGIBILITY:
Inclusion Criteria:

Each member of the couple must meet all of the following criteria to be eligible for inclusion in the study, and both members of the couple must be willing and eligible for the couple to enroll:

1. Able and willing to provide written informed consent in one of the study languages.
2. Able and willing to complete the required study procedures.
3. Currently in a heterosexual relationship (living together or not) for at least 3 months (by self-report) with the other member of the couple.
4. At time of Enrollment, expressed interest in contraception and/or HIV prevention (by self-report).

   For female partner:
5. Between the ages of 18 to 40 years (inclusive) at Enrollment, verified per site standard operating procedures (SOPs).
6. HIV negative (by self-report).

   For male partner:
7. Aged 18 years or older at Enrollment, verified per site SOPs.

Exclusion Criteria:

Potential participants who meet the following criteria will be excluded from the study along with their partner:

1. Has any significant medical condition or other condition that, in the opinion of the Investigator of Record (IoR)/designee, would preclude informed consent, make study participation unsafe (including risk for IPV as a result of study participation), complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The MTN-045 study population will consist of approximately 400 heterosexual sub-Saharan African couples of reproductive age who have been in a relationship for ≥ 3 months and are interested in contraception and/or HIV prevention. Women who are currently using contraceptives as well as those not using contraceptives will be eligible. Couples who are living together as well as those not living together will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Attributes of a DPP product that influence preferences among heterosexual couples | 12-15 months during Q2 2019/Q4 2020
  Survey questionnaires
Differences in DPP product attribute preferences when comparing individual to couples' choices (e.g., woman's individual preferences vs. preferences indicated through the joint couples decision task) | 12-15 months during Q2 2019/Q4 2020
  Discrete-Choice Experiments (DCE)

SECONDARY OUTCOMES:
Salient relationship-based and decision-making factors that influence DPP product interest and preferences | 12-15 months during Q2 2019/Q4 2020
  Survey questionnaires
Differences in attributes salient to preferences by sociodemographic factors such as age and parity that may reflect lifecourse stage | 12-15 months during Q2 2019/Q4 2020
  Survey questionnaires

OTHER OUTCOMES:
Salient relationship characteristics, norms and communication factors that influenced participants' decision-making process | 12-15 months during Q2 2019/Q4 2020
  Survey questionnaires
Differences in product preferences, when comparing individual to couples' choices, that characterize the male partner's role in females' preferences | 12-15 months during Q2 2019/Q4 2020
  Discrete-Choice Experiments (DCE)
Likelihood of using each DPP product, overall and by subgroup, as estimated through analysis of DCE data | 12-15 months during Q2 2019/Q4 2020
  Discrete-Choice Experiments (DCE)

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Minnis, PhD, Study Chair — Research Triangle Institute (RTI) International
Locations (2):
- Makerere University - Johns Hopkins University (MU-JHU) Research, Kampala, Uganda
- Zengeza Clinical Research Site, Harare, Zimbabwe

REFERENCES:
- [Result] Minnis AM, Etima J, Musara P, Browne EN, Mutero P, Kemigisha D, Mgodi NM, Nakabiito C, Shapley-Quinn MK, Stoner MCD, Hartmann M, Macagna N, Piper J, van der Straten A. Couples' Preferences for "2 in 1" Multipurpose Prevention Technologies to Prevent Both HIV and Pregnancy: Results of a Discrete Choice Experiment in Uganda and Zimbabwe. AIDS Behav. 2022 Dec;26(12):3848-3861. doi: 10.1007/s10461-022-03713-6. PMID 35674885